CLINICAL TRIAL: NCT00657137
Title: A Phase 2 Study of the Efficacy and Safety of Apricoxib in Combination With Lapatinib and Capecitabine in the Treatment of Patients With HER2/Neu+ Breast Cancer Who Have Failed Trastuzumab and Chemotherapy Including a Taxane
Brief Title: APRiCOT-B: Study to Evaluate Apricoxib in Combination With Lapatinib and Capecitabine in the Treatment of HER2/Neu+ Breast Cancer (TP2001-202)
Acronym: APRiCOT-B
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Tragara Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP2001-202; APRiCOT-B
Record Dates: First submitted 2008-03-31; First posted 2008-04-14 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: HER2/neu positive; locally advanced or metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — apricoxib; Lapatinib; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): apricoxib + lapatinib + capecitabine
  Interventions: Drug: apricoxib + lapatinib + capecitabine
- B (Placebo Comparator): placebo + lapatinib + capecitabine
  Interventions: Drug: placebo + lapatinib + capecitabine

INTERVENTIONS:
Drug: apricoxib + lapatinib + capecitabine — apricoxib: 100 mg tablets, 400 mg/day
  lapatinib: per package insert
  capecitabine: per package insert
  Arms: A
Drug: placebo + lapatinib + capecitabine — placebo: 100 mg tablets, 400 mg/day
  lapatinib: per package insert
  capecitabine: per package insert
  Arms: B

SUMMARY:
This study will compare the anti-tumor efficacy of apricoxib and lapatinib/capecitabine with placebo and lapatinib/capecitabine as measured by time to disease progression and evaluate urinary PGE-M measurements or baseline COX-2 expression in tumor tissue by IHC as a surrogate selection criterion for patients who will benefit from future treatment with apricoxib.

ELIGIBILITY:
Inclusion Criteria:

* Females with pathologically determined locally advanced or metastatic human epidermal growth factor receptor 2 positive (HER2/neu+) breast cancer
* Have progressed after treatment with chemotherapy including a taxane and trastuzumab
* Must have measurable disease by RECIST
* ECOG PS of 0,1, or 2
* MUGA scan or echocardiogram results show left ventricular ejection fraction greater than or equal to 50%

Exclusion Criteria:

* Radiation therapy within 2 weeks, chemotherapy within 3 weeks, or noncytoxic investigational agents within 4 weeks of initiating study treatment
* Evidence of New York Heart Association class III or greater cardiac disease
* History of MI, stroke, ventricular arrhythmia, or symptomatic conduction abnormality
* History of congenital QT prolongation
* Concurrent severe or uncontrolled medical disease
* Symptomatic central nervous system metastases
* Pregnant or nursing women
* Hypersensitivity or intolerance to apricoxib, lapatinib, capecitabine, 5-FU, sulfonamides, aspirin, or NSAIDs
* Severe renal insufficiency
* History of upper GI bleeding, ulceration, or perforation- Concurrent use of potent CYP3A4 inhibitors and CYP3A4 inducers
* Prior treatment with capecitabine
* Patients on anti-arrhythmic treatment
* Prior lapatinib therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine the anti-tumor activity of the combination of apricoxib/lapatinib-capecitabine compared with placebo/lapatinib-capecitabine as measured by time to disease progression. | Time to disease progression

SECONDARY OUTCOMES:
Progression-free survival and safety/tolerability | Time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Sara Zaknoen, M.D., Study Director — Tragara Pharmaceuticals, Inc.
Locations (44):
- United States (44):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Bay Area Cancer Research Group, LLC, Concord, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - Wilshire Oncology Medical Group Inc, Inland Valleys/Pomona, California
  - UCLA, Los Angeles, California
  - Olive View- UCLA Medical Center, Olive View, California
  - Cancer Care Associates Medical Group Inc, Redondo Beach, California
  - North America Research Institute, San Dimas, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Hematology Oncology Associates, Lake Worth, Florida
  - MD Anderson Cancer Center in Orlando, Orlando, Florida
  - Suburban Hematology-Oncology Associates, Lawrenceville, Georgia
  - Warren Billhartz Cancer Center, Maryville, Illinois
  - Mid-Illinois Hematology Oncology Associates, Normal, Illinois
  - Medical Consultants PC, Muncie, Indiana
  - SJMH Cancer Center, Ann Arbor, Michigan
  - Genesys Hurley Cancer Center Institute, Flint, Michigan
  - Foote Health System, Jackson County, Michigan
  - Bresline Cancer Center at Michigan State University, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy Hospital, Port Huron, Michigan
  - St. Mary's of Michigan, Saginaw, Michigan
  - St. Francis Cancer Treatment Center, Grand Island, Nebraska
  - Warren Hospital, Phillipsburg, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - Samaritan Hematology and Oncology Consulting, Corvallis, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Associates in Hematology-Oncology PC, Upland, Pennsylvania
  - Charleston Oncology Hematology Associates, Charleston, South Carolina
  - Baptist Regional Cancer Center, Knoxville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Jabboury Foundation for Cancer Research Inc, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Fletcher Allen Healthcare Inc., Burlington, Vermont
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Peninsula Cancer Institute, Newport News, Virginia
  - Madigan Army Medical Center, Tacoma, Washington